CLINICAL TRIAL: NCT06261203
Title: Low Dose Aspirin for Prevention of Early Pregnancy Loss in Women at High Risk of Preeclampsia
Brief Title: Low Dose Aspirin for Prevention of Early Pregnancy Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hany Hosny
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: The The study's findings have the potential to clarify aspirin's role in preventing adverse pregnancy outcomes related to placental dysfunction and improve the management of women at risk of placental-mediated complications.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental Group) (Experimental): About 125 Participants in the treatment group will receive 81 mg low-dose aspirin once daily starting from the time of enrollment and continuing until the end of pregnancy
  Interventions: Drug: Aspirin
- Group B (Control Group) (Placebo Comparator): About 125 Participants will receive only the routine care of pregnancy until the end of pregnancy
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — To investigate the efficacy of low dose aspirin for prevention of early pregnancy loss in women at high risk of preeclampsia.
  Other Names: Low Dose Asprin

SUMMARY:
Preeclampsia is a pregnancy-specific, multisystem disorder affecting 3% to 8% of pregnancies and remains a significant cause of maternal and neonatal morbidity and mortality worldwide.

The World Health Organization estimates that approximately 76,000 maternal deaths annually are attributed to preeclampsia, accounting for 16% of global maternal mortality, with the majority occurring in low- and middle-income countries

DETAILED DESCRIPTION:
The pathogenesis of preeclampsia (PE) is not fully understood, but it is believed to be associated with impaired early placental development, primarily attributed to defective trophoblast invasion and remodeling of the spiral arterioles .

Various mechanisms have been proposed to contribute to the development of preeclampsia, including angiogenesis, endothelial injury, oxidative stress, and inflammation, which lead to clinical manifestations such as hypertension, proteinuria, and end organ damage .

Preeclampsia is associated with severe short- and long-term maternal and neonatal morbidities, and its occurrence is influenced by risk factors such as diabetes, hypertension, multifetal gestation, as well as the severity and timing of previous preeclampsia episodes .

While low-dose aspirin (LDA) has shown some benefit in preventing preeclampsia and fetal growth restriction when initiated before 16 weeks' gestation, there is no widely effective prophylactic therapy, and delivery remains the primary approach to prevent maternal morbidity and mortality.

Recent research has indicated that LDA intervention, following firsttrimester screening of women at risk of developing preeclampsia, can significantly reduce the occurrence of preterm PE .

As such, LDA's use is increasingly considered standard practice for women at high risk of developing preeclampsia .

Nevertheless, the potential role of low-dose aspirin in preventing early pregnancy loss in this specific high-risk population remains underexplored. Given that abnormal placentation and inflammation are associated with both early and late pregnancy losses, low-dose aspirin therapy has the potential to mitigate these complications.

However, current evidence on aspirin's efficacy in preventing early pregnancy loss is limited. Considering this, we propose a randomized, double-blind, placebocontrolled trial to investigate whether low-dose aspirin (81 mg daily) administered before 16 weeks of gestation can effectively reduce the rate of early pregnancy loss in women at high risk of developing preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Before 8 weeks gestation
* Women at high risk of preeclampsia according to Royal College of Obstetricians and Gynecologists (RCOG) (Robson et al., 2013):
* Maternal age ≥ 35 years.
* Nulliparity.
* BMI ≥ 30 kg/m2.
* Smoking of r ≥ 10 cigarettes per day.
* Previous history of small for gestational age (SGA) baby.
* Previous history of stillbirth.
* Pregnancy interval < 6 months or ≥ 60months.
* Chronic hypertension.
* Diabetes with vascular disease.
* Willingness to participate in the study and provide informed written consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Use of any anticoagulant medication (e.g., heparin, warfarin, clopidogrel)
* Use of low-dose aspirin for any indication prior to the current pregnancy
* Chronic use of NSAIDs or corticosteroids
* History of bleeding disorder or active bleeding
* Any medical condition that may contraindicate the use of low-dose aspirin (e.g., peptic ulcer disease, asthma, liver, or kidney disease)
* Multiple gestation
* Inability to provide informed consent or comply with the study requirements.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Prevention of pregnancy loss | From base line to the end of pregnancy
  To investigate the efficacy of low dose aspirin (81 mg) for prevention of early pregnancy loss in women at high risk of preeclampsia.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Sayed, Professor, Study Chair — Assiut University, Faculty of medicine, Assuit.
Locations (1):
- Assuit University hospitals, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided